CLINICAL TRIAL: NCT06843343
Title: Erector Spinae Plane Block Versus Intertransverse Process Block: a Randomized Control Trial in Healthy Volunteers
Brief Title: Dispersion Following ESP Versus ITP Blocks Using Lidocaine Study
Acronym: DEVILS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00117414
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Acute Pain, Postoperative; Regional Anesthesia Block
Keywords: Erector Spinae Plane Block; ESP Block; ESP; Intertransverse Block; ITP Block; ITP; Regional Anesthesia; Paraspinal Blocks
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane (ESP) Block (Active Comparator): Participants receive ESP Block under ultrasound guidance, with 20mL of 1.5% Lidocaine on one visit.
  Interventions: Procedure: Erector Spinae Plane Block with 1.5% Lidocaine; Drug: 1.5% Lidocaine
- Intertransverse Process Block (ITP) Block (Experimental): Participants receive ITP Block under ultrasound guidance, with 20mL of 1.5% Lidocaine on the other visit.
  Interventions: Procedure: Intertransverse Process Block with 1.5% Lidocaine; Drug: 1.5% Lidocaine

INTERVENTIONS:
Procedure: Intertransverse Process Block with 1.5% Lidocaine — For the ITP block, the needle will be advanced further into the intertransverse tissue complex between the T4 and T5 transverse processes, and local anesthetic will be injected just above the superior costotransverse ligament, under ultrasound guidance.
  Arms: Intertransverse Process Block (ITP) Block
Procedure: Erector Spinae Plane Block with 1.5% Lidocaine — The ESP block will be performed by advancing the needle to the transverse process, under ultrasound guidance, with local anesthetic injected between the erector spinae muscle and the transverse process, targeting a caudad-cephalad spread.
  Arms: Erector Spinae Plane (ESP) Block
Drug: 1.5% Lidocaine — local anesthetic to be used in either the ITP and ESP block

SUMMARY:
Regional anesthesia techniques (or nerve blocks) are used to provide sensory blockade over the chest wall. The most established technique is thoracic epidural. This provides bilateral spread but is also associated with neuraxial complications, which has led to a decrease in clinical usage. Alternative peripheral nerve block techniques, such as intercostal nerve blocks, eliminate the neuraxial complications but, in turn, require numerous injections to provide unilateral coverage. The introduction of ultrasound-guided (USG) nerve blocks has generated clinical interest in the development of novel paraspinal (non-epidural) nerve block techniques, which will provide multiple dermatomal coverage with a single injection. Two such techniques are the Erector Spinae Plane (ESP) block and the Intertransverse Process (ITP) block. The Intertransverse Process (ITP) block targets a slightly deeper plane than the Erector Spinae Plane (ESP) block and was specifically designed to address the ESP block's variable anesthetic spread. Despite its potential for more localized and precise dermatomal coverage, no prior studies have directly compared the two techniques in terms of their cutaneous distribution.

Thus, this randomized, double-blinded trial aims to compare the cutaneous distribution of both these blocks in healthy adult volunteers. To compare the dermatomal sensory block distribution, the investigators will use detailed mapping with pinprick, cold, and heat stimuli.

In addition to assessing the distribution and coverage of the ESP and ITP blocks, this study also seeks to investigate the pharmacokinetics (PK) of lidocaine in each technique. The rationale for this lies in the anatomical differences between the two blocks. Theoretically, there may be a difference in the anatomical target for both blocks, but the investigators hypothesize that there is no difference in the local anesthetic absorption. Therefore, the investigators expect similar systemic absorption, the chances of local anesthetic systemic toxicity (LAST) should be equally low, and both blocks should be similarly safe.

A total of 14-18 healthy adult volunteers will be included. There will be two different procedure days, separated by at least one week. On each day, the subjects will receive a paraspinal block, according to the randomization process. Each volunteer will undergo pre-procedure screening on the first visit. The blocks will be performed on the same side, at the same level, by the same anesthesiologist, at least one week apart. An ultrasound-guided ESP block will be administered in one day, and an ITP block on the other. The order will be randomized, and both the subject and the research team member assessing the block will be blinded. Sensory testing will be performed at baseline and 60-90 minutes after the block injections. Serial samples of blood will be drawn to analyze lidocaine PK (between 0 and 240 minutes post-block).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability and willingness to comply with the study procedures and duration requirements
* ASA physical status 1 or 2
* Age ≥ 18 years

Exclusion Criteria:

* BMI > 35kg.m2
* Use of analgesics within 24 hours before the procedure
* History of thoracic trauma or surgery
* Thoracic deformities or abnormalities that may prevent proper block performance
* Thoracic tattoos
* Systemic neuromuscular disease
* Contraindications to regional anesthesia (e.g., infection, allergy, challenging sonoanatomy)
* Other known health conditions that would affect the participant's ability to successfully complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Temperature discrimination | 60 to 90 minutes post-block
  Skin temperature assessment using gloved ice on the chest wall, to discriminate blocked vs unblock areas.
Mechanical discrimination | 60 to 90 minutes post-block
  Mechanical assessment using a neuropin (pinprick) on the chest wall, to discriminate blocked vs unblock areas.
Cutaneous distribution mapping | 60 to 90 minutes post-block
  Mapping the blocked area (using the previous temperature and mechanical assessments, demarcating lines on the skin) to provide a visual map and, to calculate the area blocked.

SECONDARY OUTCOMES:
Thermography | Baseline and 60 to 90 minutes post-block
  Infrared camera will assess skin temperature of the chest wall.
Nociceptive discrimination | Baseline and 60 to 90 minutes post-block
  Nociceptive stimuli will be delivered using controlled heat to discriminate blocked versus unblocked areas on the chest wall.
Pulmonary Function Test | Baseline and 60 to 90 minutes post-block
  Peak Flow.
Lidocaine pharmacokinetics | Basiline, 10, 20, 30, 45, 60, 90, 120 and 240 minutes post block.
  Calculate lidocaine systemic absorption (Cmax).

OTHER OUTCOMES:
Adverse Events | End of study (2 days post blocks).
  Any adverse events block-related will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mendelson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No